CLINICAL TRIAL: NCT00002322
Title: Randomized, Double-Blind, Placebo-Controlled Comparative Dose-Response Study of Two Doses of Atevirdine Mesylate (U-87201E) in Combination With Fixed Doses of Zidovudine (AZT) in HIV+ Patients
Brief Title: A Study of Different Doses of Atevirdine Mesylate Plus Zidovudine in HIV-Positive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 210A; M/3330/0018
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — atevirdine; Zidovudine

INTERVENTIONS:
Drug: Atevirdine mesylate
Drug: Zidovudine

SUMMARY:
To determine the tolerance and antiviral response of two different doses of atevirdine mesylate (U-87201E) in symptomatic HIV-positive patients with CD4 counts of 50-350 cells/mm3, who also take zidovudine (AZT).

DETAILED DESCRIPTION:
Patients are randomized to 1 of 3 treatment groups: U-87201E at 1 of 2 doses or placebo administered every 8 hours. Patients must have taken AZT for at least 3 months prior to randomization.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Primary or secondary prophylaxis for opportunistic infections.

Patients must have:

* HIV infection.
* Symptoms (currently or prior to enrollment) included in Category B or C of CDC classification, although THE FOLLOWING CURRENT ACUTE MEDICAL CONDITIONS ARE NOT ALLOWED:
* Cryptococcosis
* Pneumocystis carinii pneumonia
* Herpes zoster
* Histoplasmosis
* CMV
* Hepatic or renal disease
* Lymphoma.
* CD4 count 50 - 350 cells/mm3 within 14 days prior to study entry.
* Ongoing therapy with AZT at 500 - 600 mg total daily dose for at least 3 months prior to study entry.
* Consent of parent, guardian, or person with power of attorney if less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

* Intolerance to AZT.
* Current diagnosis of malignancy for which systemic therapy will be required during the study.

Concurrent Medication:

Excluded:

* Any other investigational drugs.

Prior Medication:

Excluded:

* Cytotoxic chemotherapy within 1 month prior to study entry.
* Prior U-87201E or any other non-nucleoside antiretroviral medications, including but not limited to nevirapine, TIBO R-82150 or TIBO R-82913, L-697639 or L-696229, U-90152S, or any protease inhibitors.
* Antiretroviral agents other than AZT within 3 months prior to study entry.

Required:

* AZT for at least 3 months prior to study entry. Present use of excessive alcohol or illicit drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Los Angeles County / Health Research Assoc / Drew Med Ctr, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - Davies Med Ctr, San Francisco, California
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Boston City Hosp / FGH-1, Boston, Massachusetts
  - East Orange Veterans Administration Med Ctr, East Orange, New Jersey
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Park Plaza Hosp, Houston, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Wisconsin Community - Based Research Consortium, Milwaukee, Wisconsin